CLINICAL TRIAL: NCT06346782
Title: Feasibility, Acceptability, and Preliminary Efficacy of an Internet-based Parent-child Interaction Therapy (I-PCIT) Intervention for Children With Cancer
Brief Title: Feasibility and Acceptability of Internet-based Parent-child Interaction Therapy (I-PCIT) in Pediatric Cancer
Acronym: I-PCIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins All Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00370545
Record Dates: First submitted 2024-02-19; First posted 2024-04-04 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Pediatric Cancer; Oncology; Disruptive Behavior
Keywords: Pediatric Cancer; Oncology; Parent; Parenting; Disruptive Behavior
MeSH Terms: conditions — Neoplasms; Problem Behavior

STUDY DESIGN:
Intervention Model Description: This is a pilot feasibility trial. We are using a 2:1 (intervention: waitlist control) randomized controlled design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I-PCIT (Experimental): Participants in this study arm will receive an initial intake session with a cultural formulation interview (based on the Diagnostic and Statistical Manual (DSM-V), then will receive time-limited internet-based PCIT.
  Interventions: Behavioral: Internet-Based Parent-Child Interaction Therapy
- Waitlist Control (Active Comparator): Participants in this study arm will begin the I-PCIT intervention after a waitlist of 5-6 months. The I-PCIT intervention will be parallel to that in the I-PCIT arm.
  Interventions: Behavioral: Internet-Based Parent-Child Interaction Therapy

INTERVENTIONS:
Behavioral: Internet-Based Parent-Child Interaction Therapy — I-PCIT consists of two phases. The first phase is designed to enhance positive parent-child interactions. The second phase is designed to enhance parents' behavior management parenting behaviors.
  Other Names: I-PCIT

SUMMARY:
This study is being done to learn whether a telehealth intervention called "Internet-Based Parent Child Interaction Therapy," or I-PCIT," can help parents improve the child's behavior if the child currently or previously went through cancer treatment.

Parents who choose to be in this study will complete a survey to help researchers figure out if the parent is eligible for the larger study. If a parent is eligible for the larger study and chooses to participate, if so, the participants will be randomly assigned to either receive the I-PCIT intervention now or to be on a waitlist and begin I-PCIT in 5-6 months. The whole study consists of completing I-PCIT sessions with a clinician and completing 3-4 follow-up surveys after the initial screener survey.

DETAILED DESCRIPTION:
This study is being done to learn whether a telehealth intervention called "Internet-Based Parent Child Interaction Therapy," or I-PCIT," can help parents improve the child's behavior if the child currently or previously went through cancer treatment.

Parents who choose to be in this study will complete a survey to help researchers figure out if the parent is eligible for the larger study. If a parent is eligible for the larger study and chooses to participate, the investigators will randomly assign the participants to either receive the I-PCIT intervention now or to be on a waitlist and begin I-PCIT in 5-6 months. The whole study consists of completing I-PCIT sessions with a clinician and completing 3-4 follow-up surveys after the initial screener survey.

I-PCIT is language-dependent. The investigators will make every effort to recruit a Spanish-speaking fellow clinician for this study. However, if unable to recruit a Spanish-speaking fellow, a licensed clinical social worker and certified Spanish interpreter, will provide I-PCIT services to Spanish-speaking families. Children may participate even if the child cannot produce spoken language. Participants may request that research personnel read all assessment materials aloud in a structured interview format, in which case participants could provide verbal item responses. Because of this option, participants' ability to read and write are not requirements for participation.

The I-PCIT intervention will consist of 13 weekly telehealth sessions with a clinician who is certified in PCIT. The first telehealth session will take about 60-75 minutes. The rest of the telehealth sessions will take about 40-60 minutes. I-PCIT teaches parents how to build more positive interactions with the child and how to improve management of the child's behavior challenges.

Parents who receive I-PCIT in this study will not be charged for any I-PCIT services. Parents who are assigned to the waitlist until I-PCIT begins and may continue receiving any other services to help manage the child's behavior while waiting to start I-PCIT.

The study will last about 5-5 ½ months for parents who are assigned to start I-PCIT right away. For parents who are assigned to the waitlist to start I-PCIT in 5-6 months, parents will complete the study, including I-PCIT sessions, in about 8-9 months.

In addition to the initial survey to see if parents are eligible for I-PCIT, parents who are assigned to I-PCIT or the waitlist will also be asked to complete follow-up surveys 3-4 times during the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be parents of 2-12 year-old children who (1) currently or previously received cancer treatment and/or long-term cancer follow-up care at Johns Hopkins All Children's Hospital (JHACH).
* The child's cancer treatment must have included or plan to include chemotherapy and/or radiation.
* The child's cancer diagnosis must have been conferred at least 6 weeks prior to study enrollment. If a patient's cancer relapses during the study period, the patient's oncologist must agree to the patient continuing in this intervention.
* The parent must have access to reliable internet service (e.g., in their own home, in a friend or family member's home, via cell phone carrier) and their own smartphone, tablet, or computer to participate in telehealth intervention sessions.

Exclusion Criteria:

* Parents will be excluded if they or their child have cognitive, motor, or language delays that would preclude participation, as observed by research staff or listed in the child's medical record. Hearing impaired parents will also be excluded because I-PCIT requires the coach to verbally coach parents via bug-in-ear.
* Parents will be excluded if their child is expected to undergo bone marrow transplant (BMT) during the study or has received BMT within 2 months of study enrollment.
* The child must not be receiving end of life care, as determined by medical chart review and/or consultation with the patient's medical team.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
I-PCIT Feasibility as assessed by intervention completion | 37 weeks
  Investigators will determine I-PCIT was feasible if at least 65% of parents in the I-PCIT arm reach minimum benchmark for PCIT completion.
I-PCIT Acceptability as assessed by the Treatment Evaluation Inventory Short form | 37 weeks
  Investigators will consider I-PCIT acceptable if at least 80% of parents demonstrate scores of at least 27 on the Treatment Evaluation Inventory-Short Form. Scale range is 9 to 45. Higher scores correspond to greater acceptability of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Faith, Ph.D., Principal Investigator — Johns Hopkins All Children's Hospital
Locations (1):
- Johns Hopkins All Children's Hospital, St. Petersburg, Florida, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data will be available on request with principal investigator approval